CLINICAL TRIAL: NCT02522013
Title: Aminophylline for Patients With Post-Dural Puncture Headache: a Prospective, Multi-center, Randomized Controlled Trial
Brief Title: Aminophylline for Patients With Post-Dural Puncture Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chuanjie Wu, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAHZZU-166
Record Dates: First submitted 2015-08-08; First posted 2015-08-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Post-dural Puncture Headache
Keywords: post-dural puncture headache; Aminophylline
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Aminophylline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline group (Experimental): IV injection of aminophylline
  Interventions: Drug: Aminophylline
- isotonic saline group (Placebo Comparator): IV injection of isotonic saline group
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: Aminophylline
  Arms: Aminophylline group
Drug: isotonic saline
  Arms: isotonic saline group

SUMMARY:
Post-dural puncture headache (PDPH) is the most common complication of lumbar puncture. Its clinical manifestations are pain in the forehead and the occipital region, or diffuse headache. The pain is dull or fluctuating, becoming worse when standing and better when lying down, and is often accompanied by symptoms including a stiff neck, tinnitus, hearing loss, photophobia, and nausea, which cause great suffering to the patients1. According to epidemiological data, approximately 10% to 30% of the patients who undergo lumbar puncture suffer from PDPH within 48 hours of the procedure.Currently, commonly used treatments for PDPH include rehydration, the administration of corticotropin, caffeine, or sumatriptan, and the application of an epidural blood patch. The efficacy of theophylline has been proven in a placebo-controlled study in which 17 PDPH patients received an intravenous (IV) injection of 200 mg theophylline. The Visual Analogic Scale scores 4 hours after treatment were significantly different compared with those of the placebo group5. At present, the clinical application of theophylline has been replaced by aminophylline and doxofylline, and it is difficult to purchase theophylline in most hospitals in China and other countries.

The Aminophylline for Patients With Post-Dural Puncture Headache trial, is a prospective,randomized,double-blind,placebo-controlled trial to evaluate the efficacy and safety of an IV injection of aminophylline on post-dural puncture headache.Eligible patients were randomized in a blinded fashion(1:1) to receive IV injection of aminophyllineor or sterile isotonic saline.The investigators estimate that this trial will demonstrate that an IV injection of aminophylline could be the preferred method for the clinical treatment of PDPH.

ELIGIBILITY:
Inclusion Criteria:

* headache has developed after the dural puncture;
* PDPH was defined according to the International Classification of Headache Disorders III (ICHD-3) criteria;
* The VAS score of the headache was 5 or more than 5;
* age between 18 and 70 years old.

Exclusion Criteria:

* a previous history of headache that could interfere with PDPH diagnosis;
* a history of central nervous system diseases including intracranial hemorrhage, seizures, intracranial hypertension, and hydrocephalus;
* a history of cardiovascular system diseases including coronary heart disease, arrhythmias, and hypertension;
* a history of peptic ulcer.
* women who were pregnant, nursing, or planning a pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
pain on the Visual Analogue Scale | baseline phase
pain on the Visual Analogue Scale | 0.5 hour after the Intervention
pain on the Visual Analogue Scale | 1 hour after the Intervention
pain on the Visual Analogue Scale | 8 hours after the Intervention
pain on the Visual Analogue Scale | 1 day after the Intervention
pain on the Visual Analogue Scale | 2 days after the Intervention

SECONDARY OUTCOMES:
the overall response to treatment on the Patient Global Impression of Change | 2 days after the Intervention

OTHER OUTCOMES:
safety (occurrence of adverse reactions) | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The safety of the IV aminophylline treatment for PDPH was evaluated based on the occurrence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xue, MD, Principal Investigator — the second hospital of Hebei medcial university; Dongsheng Guan, MD, Principal Investigator — Henan Province Hospital of Traditional Chinese Medicine; Changming Wan, MD, Principal Investigator — Jingzhou Central Hospital; Zhengfei Ma, MD, Principal Investigator — Suzhou Municipal Hospital
Locations (4):
- China (4):
  - Suzhou municipal hospital, Suzhou, Anhui
  - the second hospital of Hebei medcial university, Shijiazhuang, Hebei
  - Henan Province Hospital of Traditional Chinese Medicine, Zhengzhou, Henan
  - Jinzhou central hospital, Jinzhou, Liaoning

REFERENCES:
- [Result] Feuerstein TJ, Zeides A. Theophylline relieves headache following lumbar puncture. Placebo-controlled, double-blind pilot study. Klin Wochenschr. 1986 Mar 3;64(5):216-8. doi: 10.1007/BF01711650. PMID 3517473
- [Result] Arroyo-Quiroz C, Kurth T, Cantu-Brito C, Lopez-Ridaura R, Romieu I, Lajous M. Lifetime prevalence and underdiagnosis of migraine in a population sample of Mexican women. Cephalalgia. 2014 Nov;34(13):1088-92. doi: 10.1177/0333102414529196. Epub 2014 Apr 7. PMID 24711606
- [Result] Mills MD, Hogstrom KR, Fields RS. Determination of electron beam output factors for a 20-MeV linear accelerator. Med Phys. 1985 Jul-Aug;12(4):473-6. doi: 10.1118/1.595674. PMID 3929052
- [Result] Hayallah AK, Talhouni AA, Alim AA. Design and synthesis of new 8-anilide theophylline derivatives as bronchodilators and antibacterial agents. Arch Pharm Res. 2012 Aug;35(8):1355-68. doi: 10.1007/s12272-012-0805-4. Epub 2012 Sep 1. PMID 22941478
- [Derived] Wu C, Guan D, Ren M, Ma Z, Wan C, Cui Y, Zhong P, Zhao W, Li C, Yan F, Xie J, Xue F, Lian Y, Liu H, Wang C, Ji X, Xie N. Aminophylline for treatment of postdural puncture headache: A randomized clinical trial. Neurology. 2018 Apr 24;90(17):e1523-e1529. doi: 10.1212/WNL.0000000000005351. Epub 2018 Mar 23. PMID 29572284